CLINICAL TRIAL: NCT01087840
Title: Safety, Tolerability, and Adherence to a Raltegravir-based Antiretroviral Regimen for HIV Non-occupational Postexposure Prophylaxis
Brief Title: Raltegravir Use as Nonoccupational Postexposure Prophylaxis (NPEP) in Men Who Have Sex With Men
Acronym: RAL-NPEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrew Carr (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Andrew Carr, Professor, St Vincent's Hospital
Organization: St Vincent's Hospital, Sydney (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAL-NPEP version 1.
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: HIV Prevention; HIV Infections
Keywords: HIV; nonoccupational; postexposure; prophylaxis; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir, NPEP (Experimental): Drug: Raltegravir Tablet 400mg taken orally, twice daily with or without food for 28 days along with Truvada 1 tablet taken orally daily for 28 days.
  Arms: Raltegravir/Truvada
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Drug: Raltegravir tablet 400mg is taken orally, twice daily with or without food for 28 days along with Tenofovir disoproxil fumarate/emtricitabine 300mg/200mg 1 tablet taken orally once daily with or without food for 28 days.
  Arms: Raltegravir/Truvada Other Names: Isentress/Truvada
  Other Names: Isentress; Tenofovir disoproxil fumarate/emtricitabine

SUMMARY:
The use of anti-HIV drugs following a potential sexual or injecting drug use exposure to HIV in order to try and prevent an exposure from becoming an infection is common. This is called nonoccupational postexposure prophylaxis (NPEP). The likelihood of NPEP succeeding is related to intrinsic qualities of the drugs used which includes at which point in the life cycle of the HIV virus the drugs work, how strong the drugs are against HIV, and how well tolerated the drugs are i.e. what side effects they produce. Many people skip doses during their treatment or abandon their treatment because of side effects. The anti-HIV drug raltegravir works early in the life cycle of the virus i.e. before it integrates with human DNA, is potent against HIV and causes few side effects. These qualities make it an obvious choice for use as a NPEP treatment. In this study 100 HIV negative men will receive raltegravir along with another HIV drug called truvada (commonly used in NPEP) for 28 days after a possible sexual exposure to HIV. They will be monitored closely for adverse events, side effects and for their ability to take the medicine each day for the whole 28 days. The hypothesis in this study states that raltegravir use in NPEP will be safe, well tolerated and result in a high treatment completion rate.

DETAILED DESCRIPTION:
This is a single site, 72-week, prospective, open-label, non-randomized trial. One hundred and 50 (150) eligible participants will be assigned to receive RAL 400 mg BID along with tenofovir disoproxil fumarate/emtricitabine (TVD) 1 tablet once daily (3-drug NPEP) for 28-days or TVD 1 tablet once daily (2-drug NPEP) for 28-days according to established Australian guidelines for the use of 3 or 2-drug NPEP following a potential or actual sexual exposure to HIV in men who have sex with men (MSM).1 Based on hospital NPEP data over the past 2 years, it is anticipated that 100 MSM will receive 3-drug (RAL-TVD) NPEP and 50 will receive 2-drug (TVD) NPEP. Follow-up post NPEP is for 23 weeks i.e. to week 24 post exposure.

Primary study objectives:

To describe the safety of 28 days of nonoccupational post-exposure prophylaxis(NPEP) containing raltegravir (RAL) To describe the tolerability of 28 days of NPEP containing RAL To describe on-drug adherence and regimen completion rates of 28 days of NPEP containing RAL

Secondary study objectives:

To investigate whether or not receipt of NPEP decreases, increases or has no impact on HIV risk taking behaviour To describe the effects of RAL and tenofovir disoproxil fumarate/emtricitabine (TVD) on key inflammatory biomarkers in a subset of the main study population

ELIGIBILITY:
Inclusion Criteria:

* Eligible MSM who, according to Australian NPEP guidelines, or in the opinion of the investigators, are assessed as eligible for NPEP following a potential or actual sexual exposure to HIV who present to St. Vincent's Hospital, Sydney.

Exclusion Criteria:

* Non sexual exposures
* Exposures occurring during sex between a man and a woman
* HIV infection diagnosed on baseline serological testing including indeterminate serology consistent with possible primary HIV infection
* Use of any medication contraindicated with RAL or TVD
* Serum hepatic transaminases (ALT/AST) greater than 5 times the upper limit of normal
* Serum creatinine greater than 2 times the upper limit of normal#
* Therapy with adefovir, tenofovir, emtricitabine, lamivudine, or entecavir for hepatitis B
* Baseline serological evidence of chronic/active hepatitis B
* Previous NPEP containing RAL in the study period
* A patient with a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To describe the safety of 28 days of nonoccupational post-exposure prophylaxis containing raltegravir | 28 days on drug with 5 month follow-up
  Objective AE and SAE data collection/grading utilising DAIDS data collection tool. Measurement of weight and vital signs, electrolytes, urea, creatinine, eGFR, inorganic phosphate, calcium, liver function, glucose, amylase, lipase, creatine kinase, lactate, urinalysis
To describe the tolerability of 28 days of NPEP containing raltegravir | 28 days on-drug and 5 months follow-up
  Subjective reporting of AEs with data collection/grading utilising DAIDS-AE
To describe on-drug adherence and regimen completion rates of 28 days of NPEP containing raltegravir | 28 days
  Adherence measurement by self report and pill count at 3 time points during the 28-days of NPEP

SECONDARY OUTCOMES:
To describe the context of the risk | Baseline visit day 1 of NPEP
  Context of risk event described using directed questioning around pre determined variables
To investigate whether or not receipt of NPEP decreases, increases or has no impact on future HIV risk taking behaviour | Visit 2 (day 3-5 of study), visit 7 (day 82-84 of study) visit 9 (day 166-168 of study)
  Baseline data collection of HIV risk behaviour in 6 months preceeding NPEP. Repeat data collection at week 12 and week 24 post NPEP risk event. Data collected utilising assisted completion of HIV related behaviour questionaire.
To describe the effects of raltegravir and truvada on key inflammatory biomarkers | Day 1 and day 28 of NPEP
  Measurement of CR-P, D-Dimer, IL-6 on a subset of 50 patients receiving raltegravir/truvada NPEP and a subset of 25 patients receiving truvada alone as NPEP.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fielden, RN, Principal Investigator — St Vincent's Hospital, Sydney; Anna McNulty, MBBS, FAChSHM, Principal Investigator — Sydney Sexual Health, Sydney Hospital; Phillip Read, MBBS, FAChSHM, Principal Investigator — Sydney Sexual Health, Sydney Hospital; Andrew Carr, MBBS, MD, Principal Investigator — St Vincents Hospital
Locations (2):
- Australia (2):
  - Sydney Sexual Health, Sydney Hospital, Sydney, New South Wales
  - St. Vincent's Hospital, 390 Victoria Rd, Darlinghurst, Sydney, New South Wales

REFERENCES:
- [Derived] McAllister J, Carr A. Should a protease inhibitor be standard of care for HIV postexposure prophylaxis? AIDS. 2011 Mar 13;25(5):721-2. doi: 10.1097/QAD.0b013e32834168bd. No abstract available. PMID 21368592